CLINICAL TRIAL: NCT04705532
Title: Behavioral and Neurophysiological Effects of Multichannel Executive Network tDCS Combined With Preferred Music Stimulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-280
Record Dates: First submitted 2021-01-07; First posted 2021-01-12 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Music Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS/music (Experimental): active tDCS combined with music
  Interventions: Device: tDCS; Other: Music
- sham tDCS/music (Experimental): Sham tDCS combined with music
  Interventions: Device: Sham tDCS; Other: Music
- tDCS/white noise (Experimental): active tDCS combined with white noise
  Interventions: Device: tDCS; Other: White noise
- sham tDCS/white noise (Experimental): sham tDCS combined with white noise
  Interventions: Device: Sham tDCS; Other: White noise

INTERVENTIONS:
Device: tDCS — Multi-channel tDCS will be applied over the executive network for 20 minutes at 4mA
  Arms: tDCS/music; tDCS/white noise
Device: Sham tDCS — Sham tDCS will consist of applying the same parameters as for active but the corresponding device will be turned off after 30 seconds as to simulate the initial sensation of the active current. A current of 2mA will still be used (but turned off after 30 sec). The electrodes that will be used will be the same as for the active tDCS condition and the electrodes placement as well.
  Arms: sham tDCS/music; sham tDCS/white noise
Other: Music — Subjects will listen to their preferred music for 20 minutes
  Arms: sham tDCS/music; tDCS/music
Other: White noise — Subjects will listen to a white noise for 20 minutes
  Arms: sham tDCS/white noise; tDCS/white noise

SUMMARY:
This study aims at comparing the effects of transcranial direct current stimulation combined with music on neurophysiological outcomes in healthy participants. This study also aims to evaluate the effects of tDCS combined with music on cognition.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* neurological disorders
* psychiatric disorders
* contra-indication to tDCS (eg, metallic brain implant, pacemaker)
* pregnancy
* alcool abuse
* active smoker

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
3-back | It will be measured over the course of four weeks
  The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from 3 steps earlier in the sequence.

SECONDARY OUTCOMES:
Stroop | It will be measured over the course of four weeks
  The subject has to name the font color of a printed word, while it can have a mismatch between the word and the color (ex: green is written in red).
EEG - alpha power | It will be measured over the course of four weeks
  Brain activity will be measured with an electroencephalography collected at rest. We will first look at the change in alpha power (8-12Hz)
EEG - beta power | It will be measured over the course of four weeks
  Brain activity will be measured with an electroencephalography collected at rest. We will also look at the change in other frequency bands (e.g., beta, theta, delta).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liege, Liège, Belgium